CLINICAL TRIAL: NCT05354310
Title: Vitality Oriented Innovation for the Lifecourse of the Ageing Society Intervention Study
Brief Title: The VOILA Intervention Study
Acronym: VOILA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Leiden University Medical Center (Other)
Collaborators: Maastricht University Medical Center (Other); Wageningen University and Research (Other); FrieslandCampina (Industry); ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Principal Investigator, P.Eline Slagboom, Professor of Molecular Epidemiology, Leiden University Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: NL76879.058.21
Record Dates: First submitted 2022-04-15; First posted 2022-04-29 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Aging
Keywords: Resistance Training; Nutrition; Protein supplement; Gut microbiome; Immunometabolsim; Mobility

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Active reference group (No Intervention): Only baseline measurements will be done.
- Metabolically compromised group (Experimental): Group with metabolomic mortality scores above threshold will undergo intervention. Baseline and endline measurements.
  Interventions: Combination Product: VOILA
- Mobility compromised (Experimental): Group with walking aids will undergo intervention. Baseline and endline measurements.
  Interventions: Combination Product: VOILA
- Knee replacement INT (Experimental): Group with recent knee replacement surgery will undergo intervention. Baseline and endline measurements.
  Interventions: Combination Product: VOILA
- Knee replacement Control (No Intervention): Group with recent knee replacement surgery will undergo standard care. Baseline and endline measurements.

INTERVENTIONS:
Combination Product: VOILA — Participants will be given dietary supplement powder containing protein, galactooligosaccharide (GOS), vitamin D, and calcium throughout the twelve weeks of intervention. This will be accompanied with a resistance training regime whereby participants will train three times a week for the three months. A variety of measurements will be carried out at baseline and at endline.
  Arms: Knee replacement INT; Metabolically compromised group; Mobility compromised

SUMMARY:
The multi-disciplinary and translational VOILA project presents a unique intersection between gut, immuno-metabolic, and musculoskeletal health. The main goals of the project are to develop biomarkers for healthy aging and prevent disease by maintaining quality of life in older adults. Within this umbrella project, the multimodal VOILA lifestyle intervention study will assess the impact of a twelve-week strength training and nutritional intervention in older adults with different degrees of mobility. The study will improve the current understanding of the complex relationship between gut and muscle health in different segments of mobility and obtain an insight into the heterogeneity of responsiveness between individuals.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥70 years
* A body mass index of 18.5-35.0 kg/m2
* Able to give written informed consent
* Community-dwelling
* Mentally competent with a Mini-Mental State Examination (MMSE) score of ≥24 points
* Able to follow the study protocol

Additional group-specific criteria:

Metabolically compromised group

- Framingham Risk Score ≥14 and Metabolomic Mortality Score of ≥0.173

Reduced mobility group - People able to walk but needing walking aids to walk anywhere outside their house

Total knee replacement intervention and control group

- Discharged from MUMC+ after undergoing elective knee replacement surgery (intervention starts ~4 weeks after surgery)

Active reference group

* People who meet the "Nederlandse Norm Gezond Bewegen". This means they partake in at least moderate exercise for at least 30 minutes on 5 days of the week, as determined by the SQUASH questionnaire (40).
* Framingham Risk Score of <14 and Metabolic Mortality Score of <0.173

Exclusion Criteria:

* Already using prebiotic fibres*
* Use of laxatives*
* Not willing to stop using dietary supplements in high doses (high doses: 0.10*Upper Level or more)*
* Following a structured, intense exercise programme (currently or in the last year)*
* Allergic, intolerant or hypersensitive to milk/lactose (self-reported)*
* Dietary restrictions on milk/lactose/prebiotics/vitamin D/calcium consumption*
* Abnormal hepatic or renal laboratory parameters (estimated glomerular filtration rate (eGFR) <30 ml/min/1.73 m2 (screening) or contra-indication by treating medical practitioner (data from hospital)
* Diagnosis of disorders/diseases in which a high protein intake can be harmful, such as renal impairment or failure, liver disease, or diabetes associated with nephropathy (treating medical practitioner has the decisive voice).
* Diseases, conditions or disorders which may affect the ability to follow the study protocol and which cannot be overcome with help of a caregiver Any other medical condition that may interfere with the safety of the participants during training or assessment of the outcome parameters, in the investigators' judgement
* Current participation in other scientific research that conflicts with this study (e.g. intervention studies or weight management studies)
* Not signed up to a general practitioner
* No permission to request information from the general practitioner/ treating specialist(s) about medical history, medication use.

Specific for TKR group:

* Referral to rehabilitation facility after hospital discharge
* Osteoarthritis of the knee secondary to septic arthritis, osteonecrosis, fracture, osteochondritis dissecans, or malignant processes
* Collagen disorders, e.g. Marfan and Ehler-Danlos
* Total hip prosthesis or TKR in both legs

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Muscle mass | 10 weeks
  appendicular lean mass in kg (DEXA)
Muscle function | 10 weeks
  5-times repeated chair rise test in seconds
Gut health | 10 weeks
  bifidobacteria (from stool sample) in log10 cells per gram dried faeces
Immuno-metabolic health - GLC | 10 weeks
  fasting blood glucose (GLC) in mmol/L
Immuno-metabolic health - GlycA | 10 weeks
  glycoprotein acetyls (GlycA) in mmol/L
Immuno-metabolic health - VLDL | 10 weeks
  very low-density lipoprotein (VLDL)-diameter in nm (from Nightingale 1H NMR platform)

SECONDARY OUTCOMES:
Muscle function - SPPB | 10 weeks
  Short Physical Performance Battery (SPPB)
Muscle function - TUG | 10 weeks
  Timed Up and Go test (TUG)
Muscle function - 6MWT | 10 weeks
  6-minute walking test (6MWT)
Muscle function - 1RM | 10 weeks
  1 repetition maximum test (1RM) as measured on exercise machines
Body composition - Whole body regional lean mass | 10 weeks
  DEXA whole body lean mass in kg
Body composition - Whole body regional fat mass | 10 weeks
  DEXA whole body fat mass in kg
Body composition - Regional lean mass | 10 weeks
  DEXA regional lean mass in kg
Body composition - Regional fat mass | 10 weeks
  DEXA regional fat mass in kg
Immuno-metabolic health - Hba1c | 10 weeks
  haemoglobin A1c (Hba1c)
Immuno-metabolic health - Insulin | 10 weeks
  Insulin in mol/L
Immuno-metabolic health - Blood pressure | 10 weeks
  Blood pressure in mmHg
Knee replacement group additional outcomes - CT | 10 weeks
  Single-slice CT-scans midway the upper legs
Knee replacement group additional outcomes - WOMAC | 10 weeks
  Western Ontario and McMaster Universities Arthritis Index (WOMAC).

CONTACTS AND LOCATIONS:
Overall Officials: P. Eline Slagboom, PhD, Principal Investigator — Leiden University Medical Center; Lex Verdijk, PhD, Principal Investigator — Maastricht University Medical Center; Lisette de Groot, PhD, Principal Investigator — Wageningen University & Research
Locations (3):
- Netherlands (3):
  - Wageningen University & Research, Wageningen, Gelderland
  - Maastricht University Medical Center, Maastricht, Limburg
  - Leiden University Medical Center, Leiden, South Holland

IPD SHARING:
Plan to Share IPD: Yes
Clinical data in this project will only be shared within the constraints of the informed consent. Furthermore for all permitted sharing, a data access committee (DAC) has been established in which the responsible PI of each center is present, a secretary and data manager. The data will primarily be analysed by the centers generating the data and associated partners in the VOILA project. In a later stage data access can be requested at the central contact person P.E. Slagboom (p.slagboom@lumc.nl ) and permitted by the DAC and analysed locally provided a data access agreement is signed.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Length is not determined.